CLINICAL TRIAL: NCT02925494
Title: Extension Study to Evaluate the Efficacy and Safety of Elagolix in Premenopausal Women With Heavy Menstrual Bleeding Associated With Uterine Fibroids
Brief Title: An Extension Study to Evaluate the Efficacy and Safety of Elagolix in Premenopausal Women With Heavy Menstrual Bleeding Associated With Uterine Fibroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M12-816
Record Dates: First submitted 2016-09-24; First posted 2016-10-06 (Estimated); Results first posted 2020-06-30 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Uterine Fibroids; Heavy Menstrual Bleeding
Keywords: Uterine Fibroids; Elagolix; Heavy Menstrual Bleeding; Elagolix Sodium; Elagolix plus Norethindrone Acetate
MeSH Terms: conditions — Leiomyoma; Menorrhagia | interventions — estradiol, norethindrone drug combination; elagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elagolix plus Estradiol/Norethindrone Acetate (E2/NETA) (Experimental): Elagolix 300 mg twice daily (BID) and E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) once daily (QD)
  Interventions: Drug: Estradiol/Norethindrone Acetate; Drug: Elagolix
- Elagolix (Experimental): Elagolix 300 mg BID and placebo for E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) QD
  Interventions: Drug: Elagolix

INTERVENTIONS:
Drug: Estradiol/Norethindrone Acetate — capsules
  Arms: Elagolix plus Estradiol/Norethindrone Acetate (E2/NETA)
Drug: Elagolix — film-coated tablets
  Other Names: ABT-620; elagolix sodium

SUMMARY:
This is an extension study for women who have already received six months of treatment in the phase III clinical trial M12-815 (NCT02654054) or M12-817 (NCT02691494), and will evaluate the long-term efficacy and safety of elagolix administered alone and in combination with estradiol/norethindrone acetate for an additional six months in the treatment of heavy menstrual bleeding associated with uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* Participant has completed the 6-Month Treatment Period of their respective Pivotal Study (either Study M12-815 or Study M12-817).
* Participant did not meet removal criteria in bone mineral density (BMD) decrease in the spine, total hip and femoral neck at Month 6 of the Treatment Period of their respective Pivotal Study
* Participant has negative urine and/or serum pregnancy test(s) results were consistently negative during the Treatment Period of their respective Pivotal Study and prior to first dose in this study.
* Participant's endometrial biopsy from the Month 6 Visit of their respective Pivotal Study shows no clinically significant endometrial pathology.

Exclusion Criteria:

* Participant met criteria for removal from therapy in her respective Pivotal Study.
* Participant is planning a pregnancy within the next 18 months.
* Participant has current suicidal markers as noted at the Month 6 visit of her respective pivotal study.
* Participant has any new medical conditions that may be unsuitable for participation.
* Participant is using any systemic corticosteroids for over 14 days or is likely to require treatment with systemic corticosteroids during the course of the study. Over-the-counter and prescription topical, inhaled, intranasal or injectable (for occasional use) corticosteroids are allowed.

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 433 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2019-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (124):
- United States (121):
  - Alabama Clinical Therapeutics, LLC /ID# 153217, Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC /ID# 153336, Birmingham, Alabama
  - Choice Research, LLC /ID# 153492, Dothan, Alabama
  - Brown, Pearson, Guepet Gynecology /ID# 153278, Fairhope, Alabama
  - University of South Alabama /ID# 153415, Mobile, Alabama
  - Mobile, Ob-Gyn, P.C. /ID# 153442, Mobile, Alabama
  - Mesa Obstetricians and Gynecol /ID# 153269, Mesa, Arizona
  - Core Healthcare Group /ID# 153282, Cerritos, California
  - Diagnamics Inc. /ID# 153347, Encinitas, California
  - Grossmont Ctr Clin Research /ID# 153324, La Mesa, California
  - Futura Research, Inc. /ID# 153345, Norwalk, California
  - Farid Yasharpour MD Medical Co /ID# 153482, San Fernando, California
  - Advanced Women's Health Institution /ID# 153401, Greenwood Village, Colorado
  - Medstar Health Research Institute /ID# 153321, Washington D.C., District of Columbia
  - Emerson Clinical Research Inst /ID# 162755, Washington D.C., District of Columbia
  - James A. Simon, MD, PC /ID# 153323, Washington D.C., District of Columbia
  - Helix Biomedics, LLC /ID# 153440, Boynton Beach, Florida
  - Brandon Premier Health Care, PA /ID# 165791, Brandon, Florida
  - Florida Fertility Institute /ID# 153308, Clearwater, Florida
  - Omega Research Consultants, LLC /ID# 153381, DeBary, Florida
  - KO Clinical Research, LLC /ID# 153198, Fort Lauderdale, Florida
  - Clinical Physiology Assoc. /ID# 153444, Fort Myers, Florida
  - Solutions Through Adv Rch /ID# 153283, Jacksonville, Florida
  - Meridien Research /ID# 153310, Kenneth City, Florida
  - Altus Research, Inc /ID# 153307, Lake Worth, Florida
  - South Florida Wellness & Clinic /ID# 153420, Margate, Florida
  - LCC Medical Research Institute /ID# 153296, Miami, Florida
  - Invictus Clinical Research Group,LLC /ID# 153196, Miami, Florida
  - Healthcare Clinical Data, Inc /ID# 153425, Miami, Florida
  - Ocean Blue Med Research Ctr /ID# 153225, Miami, Florida
  - Precision Research Org, LLC /ID# 153276, Miami Lakes, Florida
  - Suncoast Clinical Research /ID# 153206, New Port Richey, Florida
  - Advanced Research Institute /ID# 153413, New Port Richey, Florida
  - Clinical Associates of Orlando /ID# 153427, Orlando, Florida
  - Unified Womens Clin Research /ID# 153229, Panama City, Florida
  - All Wmns HC of West Broward /ID# 153434, Plantation, Florida
  - Oncova Clinical Research, Inc. /ID# 153497, Saint Cloud, Florida
  - Physician Care Clin. Res., LLC /ID# 153210, Sarasota, Florida
  - Qps-Mra, Llc /Id# 153456, South Miami, Florida
  - University of South Florida /ID# 153271, Tampa, Florida
  - Axcess Medical Research /ID# 153500, Wellington, Florida
  - Virtus Research Consultant,LLC /ID# 153398, Wellington, Florida
  - Comprehensive Clinical Trials /ID# 153350, West Palm Beach, Florida
  - Atlanta Medical Research Insti /ID# 153298, Alpharetta, Georgia
  - Paramount Research Solutions /ID# 153424, Alpharetta, Georgia
  - Paramount Research Solutions /ID# 160974, Alpharetta, Georgia
  - Mount Vernon Clinical Res, LLC /ID# 153403, Atlanta, Georgia
  - Atlanta Women's Research Inst /ID# 153212, Atlanta, Georgia
  - Masters of Clinical Research, Inc. /ID# 153295, Augusta, Georgia
  - Paramount Research Solutions /ID# 153351, College Park, Georgia
  - Fellows Research Alliance, Inc /ID# 153227, Savannah, Georgia
  - Clinical Research Consultants of Atlanta /ID# 153285, Suwanee, Georgia
  - Atlanta Gynecology Research Institute /ID# 200074, Suwanee, Georgia
  - Sonora Clinical Research /ID# 153231, Meridian, Idaho
  - Affinity Clinical Research /ID# 153417, Oak Brook, Illinois
  - Bluegrass Clinical Research /ID# 153280, Louisville, Kentucky
  - Clinical Trials Management, LLC - Covington /ID# 153211, Covington, Louisiana
  - Clinical Trials Management, LLC - Covington /ID# 153439, Covington, Louisiana
  - Ochsner Baptist Medical Center /ID# 153459, New Orleans, Louisiana
  - Omni Fertility and Laser Insti /ID# 153228, Shreveport, Louisiana
  - Baltimore Suburban Health /ID# 168386, Baltimore, Maryland
  - NECCR Fall River LLC /ID# 153274, Fall River, Massachusetts
  - Genesis Clinical Research /ID# 153379, Fall River, Massachusetts
  - Great Lakes Research Group,Inc /ID# 153302, Bay City, Michigan
  - Saginaw Valley Med Res Group /ID# 153498, Saginaw, Michigan
  - Wayne State University Physician Group - Southfield /ID# 153418, Southfield, Michigan
  - Accent Clinical Trials /ID# 153474, Las Vegas, Nevada
  - Office of Edmond E. Pack, MD /ID# 153411, Las Vegas, Nevada
  - Mabey, Las Vegas, NV /ID# 153314, Las Vegas, Nevada
  - Lawrence OB/GYN /ID# 153218, Lawrenceville, New Jersey
  - Jersey Shore University Medical Center /ID# 153495, Neptune City, New Jersey
  - Bosque Women's Care /ID# 153223, Albuquerque, New Mexico
  - SUNY Downstate Medical Center /ID# 153344, Brooklyn, New York
  - Manhattan Medical Research /ID# 153386, New York, New York
  - Weill Cornell Medicine /ID# 153275, New York, New York
  - Cwrwc /Id# 153313, Durham, North Carolina
  - Unified Women's Clinical Research-Greensboro /ID# 153499, Greensboro, North Carolina
  - Pinewest Ob-Gyn, Inc. /ID# 153197, High Point, North Carolina
  - Eastern Carolina Women's Centr /ID# 153341, New Bern, North Carolina
  - Unified Women's Clinical Resea /ID# 153312, Raleigh, North Carolina
  - Wake Research Associates, LLC /ID# 153402, Raleigh, North Carolina
  - Unified Women's Clinical Resea /ID# 153297, Winston-Salem, North Carolina
  - Clinical Inquest Center Ltd /ID# 153436, Beavercreek, Ohio
  - CTI Clinical Research Center /ID# 153201, Cincinnati, Ohio
  - University Hospitals Cleveland /ID# 153450, Cleveland, Ohio
  - University of Toledo /ID# 153409, Toledo, Ohio
  - Comprehensive Womens Care /ID# 153396, Westerville, Ohio
  - Legacy Medical Group-Portland /ID# 168286, Portland, Oregon
  - Main Line Fertility Center /ID# 153410, Bryn Mawr, Pennsylvania
  - Penn State University and Milton S. Hershey Medical Center /ID# 153443, Hershey, Pennsylvania
  - University of Pennsylvania /ID# 153203, Philadelphia, Pennsylvania
  - Thomas Jefferson University /ID# 153319, Philadelphia, Pennsylvania
  - Clinical Research of Philadelphia, LLC /ID# 153279, Philadelphia, Pennsylvania
  - Reading Hosp Clncl Trials Ofc /ID# 153475, West Reading, Pennsylvania
  - Medical University of South Carolina /ID# 153325, Charleston, South Carolina
  - Vista Clinical Research /ID# 153399, Columbia, South Carolina
  - Chattanooga Medical Research /ID# 153405, Chattanooga, Tennessee
  - WR-ClinSearch /ID# 153404, Chattanooga, Tennessee
  - Research Memphis Associates, LLC /ID# 153322, Memphis, Tennessee
  - Women's Health Trials /ID# 153426, Menphis, Tennessee
  - Access Clinical Trials, Inc. /ID# 153441, Nashville, Tennessee
  - Lotus Gynecology /ID# 153476, Austin, Texas
  - Texas Health Presbyterian Hosp /ID# 153339, Dallas, Texas
  - UT Southwestern Medical Center /ID# 153400, Dallas, Texas
  - Baylor Scott & White /ID# 153273, Fort Worth, Texas
  - Willowbend Health and Wellness /ID# 153458, Frisco, Texas
  - Advances in Health, Inc. /ID# 153414, Houston, Texas
  - The Woman's Hospital of Texas /ID# 153270, Houston, Texas
  - FMC Science /ID# 153289, Lampasas, Texas
  - Clinical Trials of Texas,Inc. /ID# 153209, San Antonio, Texas
  - Discovery Clinical Trials-San Antonio /ID# 153315, San Antonio, Texas
  - Houston Ctr for Clin Research /ID# 153221, Sugar Land, Texas
  - Center of Reproductive Medicin /ID# 153320, Webster, Texas
  - Tidewater Physicians for Women /ID# 153432, Norfolk, Virginia
  - Eastern Virginia Med School /ID# 153380, Norfolk, Virginia
  - Clinical Research Partners, LL /ID# 153412, North Chesterfield, Virginia
  - Clinical Research Partners, LLC /ID# 153343, Richmond, Virginia
  - Clinical Trials Virginia, Inc. /ID# 153419, Richmond, Virginia
  - Emerson Clinical Research Inst /ID# 153416, Vienna, Virginia
  - Virginia Mason Medical Center /ID# 153342, Seattle, Washington
  - Seattle Women's Health, Research, Gynecology /ID# 153306, Seattle, Washington
- Victory Reproductive Care /ID# 153299, Windsor, Ontario, Canada
- Puerto Rico (2):
  - Rodriguez-Ginorio, San Juan /ID# 153328, San Juan
  - School of Medicine University of Puerto Rico-Medical Sciences Campus /ID# 153329, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Background] Simon JA, Al-Hendy A, Archer DF, Barnhart KT, Bradley LD, Carr BR, Dayspring T, Feinberg EC, Gillispie V, Hurtado S, Kim J, Liu R, Owens CD, Muneyyirci-Delale O, Wang A, Watts NB, Schlaff WD. Elagolix Treatment for Up to 12 Months in Women With Heavy Menstrual Bleeding and Uterine Leiomyomas. Obstet Gynecol. 2020 Jun;135(6):1313-1326. doi: 10.1097/AOG.0000000000003869. PMID 32459423
- [Derived] Beck D, Winzenborg I, Liu M, Degner J, Mostafa NM, Noertersheuser P, Shebley M. Population Pharmacokinetics of Elagolix in Combination with Low-Dose Estradiol/Norethindrone Acetate in Women with Uterine Fibroids. Clin Pharmacokinet. 2022 Apr;61(4):577-587. doi: 10.1007/s40262-021-01096-w. Epub 2021 Dec 8. PMID 34878624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 433 participants who completed the 6-month Treatment Period in pivotal studies M12-815 (NCT02654054) or M12-817 (NCT02691494) were enrolled in this extension study at 114 sites in 2 countries (US [including Puerto Rico] and Canada).
Pre-assignment Details: A total of 433 participants were treated in this extension study and were grouped according to the treatment assignments in pivotal studies M12-815 and M12-817 and this extension study.
Groups:
- Placebo->Elagolix: Placebo in pivotal study and elagolix 300 mg twice daily (BID) in extension study.
- Placebo->Elagolix + E2/NETA: Placebo in pivotal study and elagolix 300 mg BID plus E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) once daily (QD) in extension study.
- Elagolix->Elagolix: Elagolix 300 mg BID in pivotal study and elagolix 300 mg BID in extension study.
- Elagolix + E2/NETA->Elagolix + E2/NETA: Elagolix 300 mg BID plus E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) QD in pivotal study and elagolix 300 mg BID plus E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) QD in extension study.
Period: Treatment Period
Arm/Group | Placebo->Elagolix | Placebo->Elagolix + E2/NETA | Elagolix->Elagolix | Elagolix + E2/NETA->Elagolix + E2/NETA
Started | 59 | 58 | 98 | 218
Completed | 50 | 43 | 79 | 182
Not Completed | 9 | 15 | 19 | 36
Period: Post-Treatment Follow-Up Period
Arm/Group | Placebo->Elagolix | Placebo->Elagolix + E2/NETA | Elagolix->Elagolix | Elagolix + E2/NETA->Elagolix + E2/NETA
Started (Completed or prematurely discontinued the Treatment Period and entered the follow-up period.) | 54 | 47 | 88 | 184
Completed | 40 | 37 | 64 | 134
Not Completed | 14 | 10 | 24 | 50
Not completed — Withdrawal by Subject | 8 | 2 | 8 | 23
Not completed — Lost to Follow-up | 3 | 2 | 9 | 10
Not completed — Other | 1 | 4 | 3 | 6
Not completed — Required Surgery/ Invasive Intervention | 1 | 2 | 2 | 6
Not completed — Pregnancy | 1 | 0 | 1 | 2
Not completed — Non-Compliance | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo->Elagolix: Placebo in pivotal study and elagolix 300 mg BID in extension study.
- Placebo->Elagolix + E2/NETA: Placebo in pivotal study and elagolix 300 mg BID plus E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) QD in extension study.
- Total: Total of all reporting groups
Arm/Group | Placebo->Elagolix | Placebo->Elagolix + E2/NETA | Elagolix->Elagolix | Elagolix + E2/NETA->Elagolix + E2/NETA | Total
Number analyzed (Participants) | 59 | 58 | 98 | 218 | 433
Age, Customized [Count of Participants; unit: Participants]
  25 to < 30 years | 0 | 3 | 1 | 4 | 8
  30 to < 35 years | 4 | 2 | 7 | 19 | 32
  35 to < 40 years | 12 | 10 | 18 | 34 | 74
  40 to < 45 years | 20 | 21 | 36 | 74 | 151
  45 to < 50 years | 16 | 16 | 30 | 77 | 139
  >= 50 years | 7 | 6 | 6 | 10 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 58 | 98 | 218 | 433
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 9 | 33 | 56
  Not Hispanic or Latino | 52 | 51 | 89 | 185 | 377
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 2
  Asian | 2 | 0 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 43 | 39 | 70 | 146 | 298
  White | 13 | 19 | 25 | 65 | 122
  More than one race | 1 | 0 | 1 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting the Criteria for Responder
Description: Percentage of responders, defined as participants who met the following conditions:
  * Menstrual blood loss (MBL) volume < 80 mL during the Final Month (the last 28 days prior to and including the last dose date), and
  * ≥ 50% reduction in MBL volume from Baseline to the Final Month.
  Participants who prematurely discontinued study drug due to "lack of efficacy," "requires surgery or invasive intervention for treatment of uterine fibroids," or "adverse events" were considered non-responders regardless of whether she meets the two aforementioned responder criteria or not.
Time Frame: From Month 0 (Baseline in Pivotal Study) to Final Month of Treatment Period (up through Month 6 in Extension Study)
Population: All participants who received at least 1 dose of study drug and had an assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo->Elagolix | Placebo->Elagolix + E2/NETA | Elagolix->Elagolix | Elagolix + E2/NETA->Elagolix + E2/NETA
Number analyzed (Participants) | 56 | 54 | 94 | 206
percentage of participants | 85.7 | 66.7 | 89.4 | 87.9

2. Secondary Outcome: Change From Baseline in MBL Volume For Each 28-Day Interval and Final Month of the Treatment Period
Description: Baseline MBL volume was defined as the mean of total MBL volume from all the qualified menstrual cycles during the Screening Period of the pivotal study, in which the total MBL volume is from all validated and non-validated sanitary products and the MBL volume of validated sanitary products only (excluding non-validated sanitary products) was greater than 80 mL.
Time Frame: Month 0 (Baseline in Pivotal Study), Extension Study: Day 1 to 28, Day 29 to 56, Day 57 to 84, Day 85 to 112, Day 113 to 140, Day 141 to 168, Final Month of Treatment Period (up through Month 6)
Population: All participants who received at least 1 dose of study drug and had an assessment at given time point.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo->Elagolix | Placebo->Elagolix + E2/NETA | Elagolix->Elagolix | Elagolix + E2/NETA->Elagolix + E2/NETA
Number analyzed (Participants) | 56 | 54 | 94 | 206
mL
  Study Day 1 to 28: number analyzed (Participants) | 54 | 51 | 94 | 205
  Study Day 1 to 28 | -151.7 (184.76) | -61.7 (212.01) | -253.4 (190.07) | -186.5 (164.38)
  Study Day 29 to 56: number analyzed (Participants) | 51 | 47 | 90 | 205
  Study Day 29 to 56 | -210.9 (234.01) | -203.1 (188.15) | -249.7 (189.81) | -191.9 (166.38)
  Study Day 57 to 84: number analyzed (Participants) | 53 | 45 | 92 | 196
  Study Day 57 to 84 | -236.9 (162.33) | -209.0 (184.90) | -255.9 (175.43) | -200.6 (159.77)
  Study Day 85 to 112: number analyzed (Participants) | 51 | 45 | 85 | 188
  Study Day 85 to 112 | -235.1 (184.87) | -204.5 (177.65) | -252.0 (175.23) | -200.5 (156.85)
  Study Day 113 to 140: number analyzed (Participants) | 49 | 42 | 78 | 181
  Study Day 113 to 140 | -237.3 (234.00) | -194.5 (213.69) | -253.9 (173.50) | -192.9 (165.42)
  Study Day 141 to 168: number analyzed (Participants) | 41 | 36 | 57 | 139
  Study Day 141 to 168 | -263.8 (199.83) | -175.4 (115.43) | -279.1 (191.44) | -211.4 (165.26)
  Final Month | -256.6 (194.04) | -186.4 (138.16) | -250.3 (182.09) | -205.6 (151.55)

3. Secondary Outcome: Percent Change From Baseline in MBL Volume For Each 28-Day Interval and Final Month of the Treatment Period
Description: as for outcome 2
Time Frame: as for outcome 2
Population: All participants who received at least 1 dose of study drug and had an assessment at given time point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo->Elagolix | Placebo->Elagolix + E2/NETA | Elagolix->Elagolix | Elagolix + E2/NETA->Elagolix + E2/NETA
Number analyzed (Participants) | 56 | 54 | 94 | 206
percentage change
  Study Day 1 to 28: number analyzed (Participants) | 54 | 51 | 94 | 205
  Study Day 1 to 28 | -46.5 (66.57) | -28.2 (72.69) | -94.0 (24.90) | -87.7 (36.24)
  Study Day 29 to 56: number analyzed (Participants) | 51 | 47 | 90 | 205
  Study Day 29 to 56 | -87.2 (46.33) | -79.4 (41.80) | -93.3 (28.77) | -87.8 (43.17)
  Study Day 57 to 84: number analyzed (Participants) | 53 | 45 | 92 | 196
  Study Day 57 to 84 | -89.9 (37.62) | -82.9 (34.79) | -96.9 (16.88) | -90.6 (32.60)
  Study Day 85 to 112: number analyzed (Participants) | 51 | 45 | 85 | 188
  Study Day 85 to 112 | -90.3 (30.26) | -82.7 (32.76) | -95.2 (19.38) | -91.2 (28.42)
  Study Day 113 to 140: number analyzed (Participants) | 49 | 42 | 78 | 181
  Study Day 113 to 140 | -90.0 (40.38) | -75.0 (65.97) | -97.7 (13.01) | -87.5 (40.67)
  Study Day 141 to 168: number analyzed (Participants) | 41 | 36 | 57 | 139
  Study Day 141 to 168 | -91.8 (30.77) | -79.3 (32.25) | -99.2 (4.31) | -89.7 (36.67)
  Final Month | -91.0 (28.74) | -78.5 (36.76) | -96.6 (18.29) | -90.8 (33.01)

4. Secondary Outcome: Percentage of Participants With Suppression of Bleeding at the Final Month
Description: Suppression of bleeding is defined as having 0 days of bleeding (spotting is allowed) during the Final Month with the interval starting from Study Day 11.
Time Frame: Final Month of Treatment Period (up through Month 6)
Population: All participants who received at least 1 dose of study drug and had an assessment.
Measure: Number; unit: percentage of participants
Groups:
- Elagolix->Elagolix + E2/NETA: Elagolix 300 mg BID plus E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) QD in pivotal study and elagolix 300 mg BID plus E2/NETA (estradiol 1.0 mg/norethindrone acetate 0.5 mg) QD in extension study.
Arm/Group | Placebo->Elagolix | Placebo->Elagolix + E2/NETA | Elagolix->Elagolix | Elagolix->Elagolix + E2/NETA
Number analyzed (Participants) | 53 | 50 | 93 | 206
percentage of participants | 88.7 | 56.0 | 89.2 | 74.8

5. Secondary Outcome: Percentage of Participants With Baseline Hemoglobin Concentration ≤ 10.5 g/dL and an Increase From Baseline > 2 g/dL at Month 6 During the Treatment Period
Time Frame: Month 6
Population: All participants who received at least 1 dose of study drug, had a baseline hemoglobin concentration of <= 10.5 g/dL and had an assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo->Elagolix | Placebo->Elagolix + E2/NETA | Elagolix->Elagolix | Elagolix + E2/NETA->Elagolix + E2/NETA
Number analyzed (Participants) | 17 | 11 | 28 | 51
percentage of participants | 70.6 | 36.4 | 71.4 | 72.5

ADVERSE EVENTS:
Time Frame: From the first dose date in Study M12-816 through up to 30 days after the last dose date. Mean (SD) treatment exposure in M12-816 was 153.7 (44.55), 145.0 (49.00), 156.5 (36.27) and 157.6 (36.11) days for the Placebo->Elagolix, Placebo->Elagolix + E2/NETA, Elagolix->Elagolix, and Elagolix + E2/NETA->Elagolix + E2/NETA arms, respectively
Description: Treatment-emergent adverse events are presented.
Arm/Group | Placebo->Elagolix | Placebo->Elagolix + E2/NETA | Elagolix->Elagolix | Elagolix + E2/NETA->Elagolix + E2/NETA
All-Cause Mortality (participants affected / at risk) | 0/59 | 1/58 | 0/98 | 0/218
Serious Adverse Events (participants affected / at risk) | 1/59 | 3/58 | 2/98 | 6/218
Other Adverse Events (participants affected / at risk) | 38/59 | 26/58 | 25/98 | 50/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo->Elagolix (N=59) | Placebo->Elagolix + E2/NETA (N=58) | Elagolix->Elagolix (N=98) | Elagolix + E2/NETA->Elagolix + E2/NETA (N=218)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PILONIDAL CYST (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OBESITY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BREAST CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FACIAL PARALYSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
METRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYSTERECTOMY (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo->Elagolix (N=59) | Placebo->Elagolix + E2/NETA (N=58) | Elagolix->Elagolix (N=98) | Elagolix + E2/NETA->Elagolix + E2/NETA (N=218)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 5 (5) | 3 (3) | 2 (2) | 9 (10)
NASOPHARYNGITIS (Infections and infestations) | 1 (2) | 1 (1) | 5 (5) | 9 (11)
TOOTH INFECTION (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 3 (3) | 4 (4) | 5 (5)
BONE DENSITY DECREASED (Investigations) | 2 (2) | 2 (2) | 6 (6) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
HEADACHE (Nervous system disorders) | 4 (4) | 3 (3) | 4 (4) | 12 (12)
ANXIETY (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
MOOD SWINGS (Psychiatric disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
METRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 15 (16) | 4 (4) | 2 (2) | 7 (8)
HOT FLUSH (Vascular disorders) | 30 (33) | 4 (4) | 3 (3) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT02925494/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT02925494/SAP_001.pdf